CLINICAL TRIAL: NCT00091091
Title: Health-Related Outcomes For Hodgkin's Disease Survivors
Brief Title: Long-Term Effects of Treatment in Patients Previously Treated for Childhood Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALTE04N1; COG-ALTE04N1 (Other: Children's Oncology Group); CDR0000383244 (Other: Clinical Trials.gov); NCI-2009-00381 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2017-02

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Children; Lymphoma
Keywords: long-term effects secondary to cancer therapy in children; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Self report/Medical record review/ clinical eval
  Interventions: Other: medical chart review; Other: questionnaire administration; Procedure: management of therapy complications

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Assessing the long-term effects of cancer treatment in cancer survivors may help improve the ability to plan effective treatment and follow-up care.

PURPOSE: This clinical trial is studying the long-term effects of treatment in patients who were previously treated for childhood Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the cumulative incidence and characterize the spectrum of selected adverse physiologic and psychosocial outcomes, using self-report and clinical evaluation, in patients previously treated for childhood Hodgkin's lymphoma.
* Compare the cumulative incidence and spectrum of self-reported adverse outcomes of these patients, using data collected at a comparable time period after diagnosis, with Hodgkin's lymphoma survivors from the Childhood Cancer Survivor Study (CCSS).
* Compare self-reported health-related outcomes with outcomes detected by clinical evaluation and medical record review of each group of patients.

OUTLINE: This is a cohort, cross-sectional, multicenter study.

* Contemporary group: Patients complete a self-report of long-term outcomes questionnaire and a comprehensive psychosocial questionnaire. A medical record review is then performed. Patients then undergo a comprehensive risk-based clinical evaluation with specific examinations and studies based upon the Children's Oncology Group Late Effects Screening Guidelines and the patients' specific therapeutic exposures.
* Childhood Cancer Survivor Study (CCSS) group: Patients undergo a telephone interview and have medical records reviewed to validate select self-reported long-term outcomes. Patient replies from the baseline CCSS questionnaire (which was completed at certain timepoints after diagnosis) are reviewed for targeted long-term outcomes.

PROJECTED ACCRUAL: Approximately 1,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Contemporary cohort

  * At least 5 years since diagnosis of Hodgkin's lymphoma

    * Diagnosed between the years 1987-2001
    * 21 and under at diagnosis
    * No evidence of disease
  * Prior treatment on 1 of the following protocols during the years 1987-2001:

    * Children's Cancer Group (CCG) CCG-5942, CCG-59704
    * Pediatric Oncology Group (POG) POG-8625, POG-8725, POG-9425, POG-9426
    * Pediatric Hodgkin's Consortium: VAMP, VEPA, VAMP/COP
    * Institutional protocols COPP/ABV, MOPP/ABVD, ABVD
* Childhood Cancer Survivor Study (CCSS) Hodgkin's lymphoma cohort

  * Current enrollment in the CCSS
  * Diagnosed between the years 1976-1986
  * Completed baseline questionnaire at comparable timepoints (as the contemporary cohort) after diagnosis

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment for primary Hodgkin disease at any one of the participating institutions 1987 - onward, or patients otherwise eligible and currently followed at one of the participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2004-12; Primary Completion 2011-06-27 (Actual)

PRIMARY OUTCOMES:
Risk for a specific adverse condition until the earliest of death, development of the adverse condition, loss to follow up, or completion of questionnaire | length of study
  The calculation of the incidence rates will be done in two ways: (a) using the self-report incidence of adverse conditions; and (b) using the incidence of adverse conditions validated by clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Debra L. Friedman, MD, MS, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (15):
- United States (15):
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin